CLINICAL TRIAL: NCT02360007
Title: Interim Buprenorphine: Leveraging Medication + Technology to Bridge Delays in Treatment Access
Acronym: IBT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Stacey C. Sigmon, Fletcher Allen Health Care, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRMS 14-063
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Opioid-related Disorders
Keywords: opioids; buprenorphine; interim treatment; opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interim Buprenorphine Treatment (Experimental): IBT participants will visit the clinic every 2 weeks while receiving the IBT package. Our integrative IBT treatment package includes five key components, each strategically chosen to maximize patient access to pharmacotherapy for opioid dependence while minimizing nonadherence, abuse and diversion: (1) Buprenorphine (BUP), (2) Computerized adherence monitoring (CAM), (3) Mobile health clinical support, (4) Urinalysis and adherence monitoring, and (5) HIV+Hepatitis Education.
  Interventions: Drug: Interim Buprenorphine Treatment (IBT)
- Waitlist Control (No Intervention): WLC participants will remain on the waitlist for their treatment of choice but complete the same scheduled follow-up assessments as IBT participants.

INTERVENTIONS:
Drug: Interim Buprenorphine Treatment (IBT) — The Interim Buprenorphine Treatment (IBT) includes:
  1. Buprenorphine (BUP)
  2. Computerized adherence monitoring (CAM): BUP will be dispensed via a portable device that makes each day's dose available only at a predetermined time.
  3. Mobile health clinical support: An Interactive Voice Response (IVR) system to deliver clinical support
  4. Urinalysis and adherence monitoring with participants contacted via IVR for random call-backs
  5. HIV+Hepatitis Education delivered via iPad
  Arms: Interim Buprenorphine Treatment

SUMMARY:
Despite the undisputed effectiveness of agonist maintenance for treating opioid dependence, current capacity is inadequate to meet need in the U.S. and internationally. Indeed, an alarming number of clinics have extensive waitlists for treatment slots. Patients can remain on these waitlists for years, placing them at elevated risk for illicit drug use, criminal activity, infectious disease, overdose and mortality during this period. These delays in treatment access represent a significant barrier to the widespread delivery of effective opioid treatment, and there is a critical need to develop creative new approaches for mitigating these delays. Our overarching goal in this application is to develop a novel Interim Buprenorphine Treatment (IBT) that can bridge delays in treatment access. Our integrative treatment package includes five key components, each strategically chosen to maximize patient access to pharmacotherapy for opioid dependence while minimizing nonadherence, abuse and diversion: Buprenorphine, Computerized adherence monitoring, mHealth clinical support delivered via Interactive Voice Response, Automated random call-backs for urinalysis and adherence monitoring, and HIV+Hepatitis Education delivered via iPad. The Primary Aim of this Stage I Behavioral and Integrative Treatment Development application is to evaluate the feasibility and initial efficacy of IBT in a 12-week randomized trial in which 70 opioid-dependent adults wait-listed for agonist maintenance are randomized to receive IBT (n=35) or continue in a Waitlist Control condition (WLC; n=35). WLC participants who have not entered treatment by Week 12 will be offered the opportunity to cross over to IBT at that time, contributing additional within-subject data with which to evaluate the efficacy of the IBT intervention. The proposed research is innovative in several important ways: By facilitating the eradication of waitlists for opioid treatment, it represents a significant departure from the status quo and stands to produce a fundamental shift in how treatment of opioid dependence is conceptualized and delivered. The IBT components are highly novel, both individually and as an integrative interim treatment package for opioid dependence. This study will be the first to investigate the utility of IBT in the patients and settings that stand to benefit most from it. The investigators also propose a multi-pronged dissemination approach that will ensure that our work is readily transported to clinical practice and will have a direct impact on real-world treatment of opioid dependence. Taken together, the proposed project will produce a highly innovative technology-assisted pharmacotherapy protocol that can be widely disseminated to increase access to life-saving opioid treatment. The overarching and specific aims of this proposal are directly relevant to NIDA's mission of improving the accessibility, implementation and effectiveness of drug abuse treatment.

DETAILED DESCRIPTION:
Agonist maintenance is the most efficacious treatment for opioid dependence. Unfortunately, demand for treatment far exceeds available capacity. An alarming number of clinics have extensive waitlists for treatment slots (Gryczynski et al., 2009; Peles et al., 2012; Peterson et al., 2010). Patients can remain on these waitlists for years, placing them at elevated risk for illicit drug use, criminal activity, infectious disease, overdose and mortality during this period (Peles et al., 2013; Warner-Smith et al., 2001; Wenger & Rosenbaum, 1994). These delays in treatment access represent a significant barrier to the widespread delivery of effective opioid treatment, particularly in rural areas where there are fewer providers and substantial unmet treatment need. One important effort to increase access has been to extend interim methadone treatment (IMT; i.e., daily methadone + emergency counseling only) to individuals awaiting enrollment into a methadone program. IMT significantly reduces illicit opioid use and criminality and increases likelihood of treatment entry (Schwartz et al., 2006, 2007, 2009a,b, 2011). However, methadone treatment in the U.S. is limited to licensed specialty clinics, it requires frequent clinic visits, and the medication itself has risks of diversion, abuse and overdose. Hence, methadone's regulatory and pharmacological features substantially constrain the ability of IMT to expand access to opioid treatment.

Our overarching goal in this application is to develop a novel Interim Buprenorphine Treatment (IBT) that can bridge delays in treatment access. Our integrative treatment package includes five key components, each strategically chosen to maximize patient access to pharmacotherapy for opioid dependence while minimizing nonadherence, abuse and diversion: (1) Buprenorphine (BUP): Due to its pharmacological profile, BUP has less risk of abuse and overdose and is available without the rigid dosing regulations required for methadone. Thus, we will use BUP in this interim-treatment model. (2) Computerized adherence monitoring (CAM): We will use CAM to promote medication adherence and reduce diversion risk. BUP doses will be dispensed via a state-of-the-art portable device that makes each day's dose available only at a predetermined time, after which all medication is inaccessible. (3) Mobile health clinical support: mHealth platforms use information and communication technology to deliver patient monitoring, education and support beyond the confines of the medical office. Interactive Voice Response (IVR) systems are especially promising in that they provide customized support via phone with low cost, consistent delivery, 24-hour availability, privacy and convenience. We will develop an IVR system to deliver clinical support with branching logic in a seamless fashion as well as immediate connection with staff or crisis service if needed. (4) Urinalysis and adherence monitoring: We will develop an automated call-back procedure to contact participants via IVR at randomly-determined intervals and notify them to return to the clinic to provide a urine specimen and present the CAM device for inspection. This component will provide a rigorous but efficient method for supporting abstinence and adherence over an extended period of lower-frequency visits. (5) HIV+Hepatitis Education: We have developed an intervention that produces significant improvements in HIV and hepatitis knowledge. However its resource-intensive in-person format may limit its utility in IBT. We will adapt our intervention for delivery via iPad, a state-of-the-art platform with portability, sophisticated functionality and widespread appeal.

The primary aim of this Stage I Behavioral and Integrative Treatment Development application is to develop a novel, manual-based IBT platform to increase access to opioid treatment. During Months 1-6 we will refine treatment components using feedback from stakeholders. During the remaining study period, we will evaluate the feasibility, acceptability and initial efficacy of IBT in a 12-week proof-of-concept trial in which 70 opioid-dependent adults wait-listed for agonist maintenance are randomized to receive IBT (n=35) or continue in a Waitlist Control condition (WLC; n=35). IBT participants will visit the clinic every 2 weeks while receiving the IBT package described above. WLC participants will remain on the waitlist for their treatment of choice but complete the same scheduled follow-up assessments as IBT participants. WLC participants who have not entered treatment by Week 12 will be offered the opportunity to cross over to IBT at that time, contributing additional within-subject data with which to evaluate the efficacy of the IBT intervention.

By facilitating the eradication of waitlists, the proposed research represents a significant departure from the status quo and stands to produce a fundamental shift in how treatment of opioid dependence is conceptualized and delivered. The IBT components are highly novel, both individually and as an integrative treatment package for opioid dependence. This study will also be the first to investigate the utility of IBT in the patients and settings that stand to benefit most from it and includes a multi-pronged dissemination plan to ensure that our findings are readily transported into real-world clinical practice. Taken together, the proposed project will produce a highly innovative technology-assisted pharmacotherapy protocol that can be widely disseminated to increase access to life-saving opioid treatment. These aims are directly relevant to NIDA's mission of improving the accessibility, implementation and effectiveness of drug abuse treatment.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the trial, participants must be >18 years old, in good health, meet DSM-IV criteria for opioid dependence, provide an opioid-positive urine and be currently waitlisted.
* To minimize disruption due to treatment becoming available during the study, we will limit enrollment to those who joined a waitlist in the prior 12 months.

Exclusion Criteria:

* Those with a significant psychiatric or medical illness that may interfere with consent or participation will be excluded, as will those who are pregnant or nursing.
* Females will be tested for pregnancy and, should a participant become pregnant during the trial, her participation will be terminated and she will be assisted with accessing treatment at the high-risk pregnancy clinic.
* Those dependent on sedative-hypnotics will be excluded, due to the medical risks and notably low success rates with sedative-dependent opioid abusers (Stitzer & Chutuape, 1999).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Illicit opioid abstinence | 12 weeks
  IBT and WLC experimental groups will be compared on percentage of subjects abstinent for illicit opioids across Week 4, 8, and 12 assessments

SECONDARY OUTCOMES:
ASI subscale scores | 12 weeks
  IBT and WLC experimental groups will be compared on ASI composite subscale scores across Week 4, 8, and 12 assessments

CONTACTS AND LOCATIONS:
Locations (1):
- Substance Abuse Treatment Center, University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Derived] Streck JM, Ochalek TA, Badger GJ, Sigmon SC. Interim buprenorphine treatment during delays to comprehensive treatment: Changes in psychiatric symptoms. Exp Clin Psychopharmacol. 2018 Aug;26(4):403-409. doi: 10.1037/pha0000199. Epub 2018 Jun 25. PMID 29939049